CLINICAL TRIAL: NCT06289894
Title: A Phase I, Open-label, Single Arm Study to Evaluate the Safety, Tolerability, and Antitumor Activity of BRY805 in Participants With Advanced Solid Tumors
Brief Title: A Study of BRY805 in Participants With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Adjustment of the company's R&D strategy
Sponsor: BioRay Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRY805-101
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BRY805 (Experimental)
  Interventions: Drug: BRY805 injection

INTERVENTIONS:
Drug: BRY805 injection — BRY805 will be administered via IV infusion every 3 weeks. , Six dose levels of 0.3, 1, 3, 9,18 and 30 mg/kg will be tested

SUMMARY:
This is a phase 1 open label multicenter study to evaluate safety, tolerance and the maximum tolerance of BRY805 administered intravenously (IV) once every three weeks in participants with advanced solid tumors, so as to confirm the recommended phase 2 dose of BRY805 and obtain the preliminary efficacy information of participants with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* 1. Willing and able to provide signed informed and to comply with all study procedures; 2. Male or female ≥ 18 years; 3. Advanced malignant solid tumor patients who have experienced treatment failure using established therapeutic methods, have no viable standard treatment options available, or are unable to tolerate standard therapy; 4. ECOG score ≤ 1; 5. Life expectancy ≥ 3 months; 6. Considering that the phase I trial mainly evaluates the safety and tolerability of the drug, subjects who cannot measure the lesion can be enrolled in the dose escalation phase to obtain more safety, pharmacokinetic and pharmacodynamic results. Enrolled subjects who may have been expanded at 1-3 doses that may have been selected in the early period, have at least one measurable lesion in the baseline period according to RECIST v1.1; 7. Recovery, to Grade 0-1, from adverse events related to prior anticancer therapy except alopecia, < Grade 2 sensory neuropathy and endocrinopathies controlled with hormone replacement therapy; 8. Sufficient organ and bone marrow function; 9. Female subjects of childbearing age must have a negative serum pregnancy test result when they enter this study (tested within 1 week before the first dose); Female subjects of childbearing potential or male subjects whose sexual partner is a female of childbearing age, who are willing to use appropriate and effective contraceptive measures such as abstinence and double barrier methods (such as condoms plus contraceptive diaphragms), oral contraceptives, intrauterine device insertion, etc., during the study period and within 6 months after the last dose.

Exclusion Criteria:

* 1. Hypersensitivity to study drug or components of its formulation; or have had a severe allergic reaction to other monoclonal antibodies; 2. Prior treatment with NKG2A-targeted agents; 3. Participants will be excluded if they meet any of the following criteria:

  * Major surgery within 4 weeks prior to the first dose, or anticipated major surgery during the study, minor surgery within 2 weeks prior to the first dose;

    * Use of immunosuppressive medications within 2 weeks prior to the first dose; nasal and inhaled corticosteroids or physiologic doses of systemic steroids (i.e., no more than 10 mg/day of prednisone or equivalent pharmacophysiological doses of other corticosteroids) are allowed in the absence of active autoimmune disease;

      * Live vaccine administration within 4 weeks prior to the first dose, at any time during the study, or within 1 month after the last dose; ④ Received anti-tumor therapy (including chemotherapy, radiotherapy, immunotherapy, endocrine therapy, targeted therapy, biological therapy, or tumor embolization) within 5 half-lives or 4 weeks (whichever is shorter) prior to the first dose, or used therapeutic radiopharmaceuticals (strontium, samarium, etc.) within 8 weeks prior to the first dose; ⑤ Participation in other clinical trials within 4 weeks prior to the first dose.

        4. Active autoimmune disease or history of autoimmune disease that may recur, including but not limited to systemic lupus erythematosus, psoriasis, rheumatoid arthritis, inflammatory bowel disease, Hashimoto's thyroiditis, etc. Except for conditions that require only alternative therapy (e.g., residual hypothyroidism due to autoimmune thyroiditis); 5. Symptomatic central nervous system metastases. Asymptomatic patients with CNS metastases who are radiographically and neurologically stable ≥for 4 weeks after CNS-directed therapy and are on stable or reduced doses of corticosteroids are eligible for study entry; 6. History of any malignancy within the past 5 years, with the exception of cured cervical carcinoma in situbasal, basal cell or squamous epithelial cell carcinoma of the skin, localized prostate cancer, ductal carcinoma in situ of the breast, or other malignancies that have been previously treated and judged by the investigator to have stable disease status; 7. Active HIV, hepatitis B or hepatitis C virus. A positive TP specific antibody test requires testing for syphilis non-specific antibodies; 8. Severe cardiovascular disease, including CVA, TIA, myocardial infarction, or unstable angina within 6 months of study entry; NYHA class III or IV heart failure within 6 months of study entry; Uncontrolled arrhythmia within 6 months of study entry; 9. QTcF interval ≥ 470 ms; 10. Uncontrolled hypertension (systolic blood pressure >160 mmHg and diastolic blood pressure >100 mmHg), a history of hypertension crisis, or a history of hypertensive encephalopathy; 11. Active infection requiring intravenous therapy within 2 weeks prior to the first dose; 12. Active tuberculosis, or anti-tuberculosis therapy within 1 year prior to screening; 13. Interstitial lung disease, such as interstitial pneumonia, pulmonary fibrosis, etc., or non-infectious pneumonia; 14. Diseases affecting intravenous infusion and venous blood collection; 15. Has bleeding tendencies or is receiving thrombolytic or anticoagulant therapy; 16. History of allogeneic organ or stem cell transplantation; 17. History of prior grade 3-4 immune-related adverse events or immune-related adverse events requiring discontinuation of treatment; 18. Has a known or suspected condition that is incapable of complying with the study protocol (such as a history of psychotropic substance abuse, alcohol dependence, psychological disorder, or drug abuse); 19. Participants considered unsuitable for inclusion or who may not be able to complete the study for other reasons by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2024-03-13 (Actual); Primary Completion 2025-05-16 (Actual); Study Completion 2025-07-04 (Actual)

PRIMARY OUTCOMES:
Occurrence of Drug Limited Toxicities (DLTs) | From Time of First dose through DLT observation period, 21 days
  To assess by the occurrence of Drug Limited Toxicities (DLTs)
Type and incidence of Treatment-emergent adverse event (TEAEs) and serious adverse events (SAEs) | From first dose until up to 91 days after the last dose
  To assess by the occurrence of Treatment-emergent adverse event (TEAEs) and serious adverse events (SAEs)

SECONDARY OUTCOMES:
BRY805 Serum Concentrations | From first dose to 31 days after the last dose
  Serum concentrations will be calculated for BRY805
Number of Participants with BRY805 Antibodies | From first dose to 31 days after the last dose
  Antibodies to BRY805 will be assessed to evaluate potential immunogenicity
Overall Response Rate (ORR) | Until study termination (approximately 2 years)
  The proportion of participants who achieved CR or PR. Disease response will be assessed by the investigator using RECIST v1.1 and immune RECIST (iRECIST).
Disease Control Rate (DCR) | Until study termination (approximately 2 years
  The proportion of participants who achieved stable disease (SD), PR, or CR
Progression-Free Survival (PFS) | Until study termination (approximately 2 years)
  The time from the first dose to the first documented PD or death due to any cause, whichever occurs first

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong Tumor hospital, Jinan, Shandong, China